CLINICAL TRIAL: NCT02268825
Title: A Phase I Study of MK-3475 in Combination With Chemotherapy and Supplemental Celecoxib in Patients With Advanced GI Cancers (Colorectal/Appendiceal Adenocarcinoma, Gastroesophageal, Pancreatic and Biliary)
Brief Title: Phase I Study MK-3475 With Chemotherapy in Patients With Advanced GI Cancers
Acronym: MK-3475 GI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Merck requested to change MK-3475 dosing schedule; PI decided to close instead
Sponsor: University of Utah (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI76239
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Advanced GI Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-3475 treatment arm, all patients (Experimental)
  Interventions: Drug: MK-3475

INTERVENTIONS:
Drug: MK-3475 — MK-3475 in combination with mFOLFOX6 in a 14 day cycle
  Phase 1 and safety expansion Phased Regimen mFOLFOX6 Administered Day 1 of each cycle Leucovorin 400 mg/m2 IV 5-FU 400 mg/m2 IV bolus followed by 2400 mg/m2 IV over 46 hrs Oxaliplatin (Eloxatin) 85 mg/m2 IV
  MK-3475 IV to be administered before mFOLFOX6 starting with Cycle 3 (after 28 days of chemotherapy alone); day 1 of each cycle (q 2 weeks)
  Phase 1: 2 dose levels of MK-3475 Level -1: 50mg IV q 2 weeks Level 1: 75mg IV q 2 weeks Level 2: 200mg IV q 2 weeks
  Safety Expansion: MK-3475 at highest tolerated dose

SUMMARY:
This is a Phase I dose escalation trial to assess MTD of MK-3475 in combination with mFOLFOX6 followed by a safety expansion open label, nonrandomized trial with MK-3475 at MTD in combination with mFOLFOX6 and supplemental celecoxib in 4 cohorts of advanced/metastatic GI malignancies (pancreatic, gastro esophageal, colorectal/appendiceal adenocarcinoma and biliary carcinoma) to assess response rate, clinical benefit rate, progression free survival and overall survival. The safety expansion cohort will assess the effect of the addition of celecoxib to patients that do not respond to combination MK-3475/mFOLFOX treatment.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Patients with any locally advanced or metastatic gastrointestinal malignancy which mFOLFOX6 is indicated for treatment
* Safety expansion: Patients with one of the following locally advanced unresectable or metastatic pathologically confirmed diagnosis: Colorectal Carcinoma and Appendiceal Adenocarcinoma, Gastro-Esophageal -Carcinoma Note: esophageal squamous cell carcinoma is exclusionary, Biliary -Tract Carcinoma Note: Hepatocellular carcinoma is excluded, Pancreatic Carcinoma
* Patients must be willing to provide and have available formalin fixed paraffin embedded tissue sample from archival tissue or newly obtained core or excisional biopsy of a tumor lesion for central analysis. Note: Fine Needle Aspiration's (FNA), frozen samples, plastic embedded samples, cell blocks, clots, bone, bone marrow, or cytologic specimens are exclusionary
* Patients must have measurable disease based on irRECIST (Safety expansion only)
* Patients must be 18 years of age on day of signing informed consent
* Have a performance status of 0 or 1 on the ECOG Performance Scale
* Patients must demonstrate adequate organ function as based on screening labs performed within 14 days of treatment initiation
* Patients are allowed to have received prior treatment with mFOLFOX6. If patients are currently receiving treatment with mFOLFOX6, the subject must have documented disease progression. Patients must also be able to tolerate standard mFOLFOX6. Reduced dosing of mFOLFOX6 at enrollment is exclusionary.
* Patients must be able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for greater than 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Note: Dexamethasone prior to treatment on day 1 of each treatment cycle is allowed
* Subjects with greater than or equal to Grade 2 neuropathy
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., greater than or equal to Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* History of greater than or equal to grade 3 allergic reaction to mFOLFOX6 (patients successfully desensitized to oxaliplatin are eligible or those willing to undergo desensitization during the first two cycles of mFOLFOX6 per institutional guidelines)
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators, topical steroids or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study
* Has history of interstitial lung disease or active, non-infectious pneumonitis requiring steroids.
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Note: testing not required at baseline unless clinically indicated
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). Note: testing not required at baseline for unless clinically indicated
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Patients are ineligible if they plan on regular use of NSAIDs at any dose more than 2 times per week (on average) or aspirin at more than 325 mg at least three times per week, on average. Low-dose aspirin not exceeding 100mg/day is permitted. Patients who agree to stop regular NSAIDS or higher dose aspirin are eligible and no wash out period is required.
* The patient has significant bleeding disorders or vasculitis. History of significant (in the opinion of the investigator) upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years. Patients with a history of ulceration, bleeding or perforation in the lower bowel are not excluded.
* Prior allergic reaction or hypersensitivity to sulfonamides (may be allowed per investigator discretion based on patient history), celecoxib or NSAIDs.
* Cardiac risk factors including: 1) Uncontrolled high blood pressure (systolic blood pressure greater than 150); 2) Unstable angina; 3) History of documented myocardial infarction or cerebrovascular accident; 4 New York Heart Association class III or IV heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Safety of combination mFOLFOX and MK-3475 | Patient safety will be evaluated throughout the treatment period (treatment with MK-3475 and FOLFOX) which is expected to last 4-6 months for each patient.
  Routine safety and tolerability will be evaluated from the results of reported signs and symptoms, scheduled physical examinations, vital sign measurements, and clinical laboratory test results. More frequent safety evaluations may be performed if clinically indicated or at the discretion of the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States